CLINICAL TRIAL: NCT00943189
Title: Fetal Anomalies Scan at the Time of Nuchal Translucency Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Liat Gindes, Sheba Medical Center
Other Study IDs: SHEBA-08-4934-LG-CTIL
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Fetal Anomalies
Keywords: Fetal anomalies scan at the time of NT study
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Purpose: Fetal anomalies scan at the time of Nuchal Translucency (NT) study.

DETAILED DESCRIPTION:
Prospective study of patients at 12-14 weeks gestation that are coming for NT examination is conducted. Meticulous ultrasound examination will be done to the fetuses using trans vaginal and transabdominal techniques. The patients will receive only the NT information. Only in cases of detection of severe fetal anomalies the patient will get the information of the examination and counseling according to the findings. All patients will be asked to provide information of the 15 weeks early comprehensive ultrasound examination. The NT examination will be compared to the 15 weeks ultrasound. All patients will be asked to give information after delivery of the baby's health condition.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women at 12-14 weeks

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All pregnant women at 12-14 weeks of gestation that are coming for nuchal translucency examination and willing to participate in the study.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2008-06

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel